CLINICAL TRIAL: NCT05050825
Title: Validation of an Assisted Medical Care Strategy Composed of a Clinical Decision Support System and RDTs to Reduce Antibiotic Prescription in Non-severe Acute Disease in Children 15 Years Old and Younger in Senegal
Brief Title: Validation of a CDSA Strategy to Reduce Antibiotic Prescription in Senegal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Institut Pasteur de Dakar (Other); Ministry of Health, Senegal (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FE007
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Malaria; Dengue; Influenza -Like Illness; Diarrhea; Pneumonia; Acute Febrile Illness
Keywords: clinical algorithms; mHealth; Integrated management for childhood illness
MeSH Terms: conditions — Malaria; Dengue; Diarrhea; Pneumonia

STUDY DESIGN:
Intervention Model Description: Control (routine practice) vs Intervention ("CDSA" strategy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSA strategy (Experimental): Children and adolescents presenting with non-severe acute febrile illness or diarrhea managed by healthcare workers trained on the CDSA strategy
  Interventions: Other: Patient clinical management based on the CDSA strategy
- Routine practice (No Intervention): Children and adolescents presenting with non-severe acute febrile illness or diarrhea managed by healthcare workers according to routine practice at the health facility

INTERVENTIONS:
Other: Patient clinical management based on the CDSA strategy — The CDSA strategy is a combination of point of care tests (rapid diagnostic tests targeting malaria, dengue fever and streptococcus group a sore through) and a mHealth tool that provides patient management recommendations, including treatment, based on an algorithm integrating patient clinical signs and symptoms, history and diagnostic test results.
  Arms: CDSA strategy

SUMMARY:
This trial aims to validate a novel clinical care strategy based on a electronic clinical decision support algorithm (CDSA) combined with point of care rapid diagnostic tests by evaluating its impact on antibiotic prescription and clinical outcome of children and adolescent presenting at primary healthcare facilities with non-severe acute illness compared to routine practice. The trial also aims to assess the usability of the CDSA strategy. The study will be conducted in primary healthcare facilities across different epidemiological regions of Senegal.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing fever or diarrhea
* ongoing fever will be defined objectively or as a reported fever, defined as : axillary temperature ≥37.5°C or tympanic, oral or rectal temperature ≥38.0°C; and fever duration ≤ 10 days
* ongoing diarrhea will be defined as at least 3 abnormal stools during the last 24hrs
* First consultation for the current illness
* Feasibility of contact between the patient (or his/her designated relative) and the study team at day 3 and day 7
* Written informed consent by the caretaker/legally acceptable representative

Exclusion Criteria:

* Infants less than 6 months of age
* Age ≥ 15 years
* Clinical status requiring immediate transfer to an appropriate care facility/ severe illness

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 470 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the CDSA strategy when compared to routine practice in terms of clinical status assessed at Day 7 | 4 months
  This will be measured as point estimates of the percent change of patient with resolved illness at Day 7 in the intervention arm, as compared to the control arm.
Superiority of the CDSA strategy when compared to routine practice in terms of antibiotic prescription at Day 0 | 4 months
  This will be measured as point estimates of the percent change of antibiotic prescription at Day 0 in the intervention arm, as compared to the control arm and to site-specific historical data. This measure aims to assess rational use of antibiotics using the CDSA strategy compared to routine practice.

SECONDARY OUTCOMES:
Antibiotic prescription rate during 7 days of follow-up in the intervention arm compared to the control arm | 4 months
  This measure will further assess rational antibiotic prescribing using the CDSA strategy compared to routine practice.
Diagnostic performance of the dengue rapid diagnostic test (RDT) | 4 months
  The performance of the dengue RDT used in health facilities will be assessed against reference standards.
Identification of risk factors associated with viral and bacterial infections | 4 months
  This measure aims to better characterize viral and bacterial infections in children and adolescents presenting with acute illness in these settings and improve the next version of the algorithm.

OTHER OUTCOMES:
Usability of the CDSA strategy | 4 months
  This measure will determine the ease of use of the CDSA strategy. This will be assessed through questionnaires administered to end users at the beginning and end of participant inclusion; the assessment of data completeness comparing historical collected-on-paper to study data; and passive collection of the platform performance indicators autogenerated by the platform.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Taieb, MD, Principal Investigator — Institut Pasteur de Dakar; Aliou Barry, MD, Principal Investigator — Institut Pasteur de Dakar
Locations (4):
- Senegal (4):
  - PS Ndiaye-Fatick, Fatick
  - PS Kedougou-Dalaba, Kédougou
  - PS Mbour-Toucouleur, Mbour
  - PS Pont-Tambacounda, Tambacounda